CLINICAL TRIAL: NCT06985836
Title: Effect of Mulligan Mobilization With or Without Niel Asher Technique on Pain, Range of Motion and Disability in Patients With Adhesive Capsulitis
Brief Title: Effect of Mulligan Mobilization With or Without Niel Asher Technique in Patients With Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0180
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; frozen shoulder; mannual therapy
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Mobilization and Niel Asher technique (Experimental): Shoulder mobilization that includes:
  * Mulligan mobilization technique for shoulder external rotation and abduction as described by Mulligan. 3 sets of 10 repetitions with 1 minute rest between sets, 3 times a week for 4 weeks are performed
  * Niel Asher technique provided for 3 sessions a week for 4 weeks
  Interventions: Other: Mulligan Mobilization and Niel Asher technique; Other: Mulligan Mobilization and Conventional physiotherapy.
- Mulligan Mobilization and Conventional physiotherapy. (Active Comparator): Group B Will receive Baseline Physical therapy treatment and mulligan mobilization.
  Standardized Physiotherapy treatment will be:
  * Modalities i.e. heating pad and TENS for ten Minutes
  * Postural correction exercises / Scapular retraction
  * Therapeutic Exercise : Codman' s, finger ladder, wand exercises
  * End Range Gleno-humeral joint stretching Both groups will come four times per week for a total of 4 weeks. Pre and post treatment values of both groups will be analyzed
  Interventions: Other: Mulligan Mobilization and Conventional physiotherapy.

INTERVENTIONS:
Other: Mulligan Mobilization and Niel Asher technique — * Mulligan mobilization technique for shoulder external rotation and abduction as described by Mulligan. 3 sets of 10 repetitions with 1 minute rest between sets, 3 times a week for 4 weeks are performed
  * Niel Asher technique provided for 3 sessions a week for 4 weeks
  Arms: Mulligan Mobilization and Niel Asher technique
Other: Mulligan Mobilization and Conventional physiotherapy. — * Modalities i.e. heating pad and TENS for ten Minutes
  * Postural correction exercises / Scapular retraction
  * Therapeutic Exercise : Codman' s, finger ladder, wand exercises
  * End Range Gleno-humeral joint stretching Both groups will come four times per week for a total of 4 weeks. Pre and post treatment values of both groups will be analyzed.

SUMMARY:
Adhesive capsulitis is a prevalent condition characterized by pain and stiffness in shoulder joint and surrounding muscles shows decrease range and strength in patients with adhesive capsulitis. This study aims to determine the effect of mulligan mobilization with or without Niel Asher technique on pain, range of motion and disability in patients with adhesive capsulitis. This study will be a randomized controlled trial and will be conducted in Ibne-siena Hospital Multan and Multicare physiotherapy clinic. Non-probability convenience sampling will be used to collect the data. Sample size of subjects with age group between 40 to 60 years will be taken. Data will be collected from the patients having present complaint of adhesive capsulitis. Outcome measures used will be Numeric pain rating scale (NPRS) for shoulder pain and SPADI for shoulder disability and Universal Goniometer (GU) for Range of motion. An informed consent will be taken. Subjects will be selected on the basis of inclusion and exclusion criteria. Subjects will be divided into two groups by random number generator table. Both the Groups will receive heating pad, TENS. Group A will receive Mulligan Mobilizations and Neil Asher technique, and Group B will receive Mulligan mobilization and Conventional Treatment. Outcome measures will be measured at baseline and after 4 weeks. Data analysis will be done by SPSS version 26.

ELIGIBILITY:
Inclusion Criteria:

* Age group 40-60 year
* Both gender male and female
* Stage 2 primary adhesive capsulitis with capsular pattern of restriction (rotation>abduction>flexion)
* Pain in shoulder should be ≤7 on NPRS
* Patient is willing to perform.

Exclusion Criteria:

* • Diabetes

  * Malignancy
  * Infection
  * Arthoplasty
  * Pregnancy
  * Neurological disorders
  * Fracture
  * Thyroid diseases

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | baseline and fourth week
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates " no pain" and 10 indicates " worst pain" . NPRS have shown high test- retest reliability (r = 0.96 and 0.95, respectively)
Universal Goniometer (UG) | baseline and fourth week
  The range of motion will be measured using universal goniometer that has an inter-rater reliability (ICC2, 2 = 0.79 to 0.92) for shoulder.
Shoulder disability and shoulder Index SPADI | baseline and fourthweek
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper- extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder. The reliability coefficient is ICC >0.89 for Shoulder.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- Ibne Siena hospital Multan., Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doner G, Guven Z, Atalay A, Celiker R. Evalution of Mulligan's technique for adhesive capsulitis of the shoulder. J Rehabil Med. 2013 Jan;45(1):87-91. doi: 10.2340/16501977-1064. PMID 23037929
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561